CLINICAL TRIAL: NCT07166822
Title: The Role of Mobile Apps in Promoting Cardiovascular Health and Motivation to Exercise During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Leryn Reynolds, Associate Professor, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FF2
Record Dates: First submitted 2025-08-27; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular (CV) Risk; Exercise
Keywords: pregnant; cardiovascular; mobile app; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm who will use the BumptUp mobile exercise app (Experimental): This group will have access to "BumptUp" mobile exercise app and will be provided with an educational brochure (Exercise during pregnancy)
  Interventions: Behavioral: Experimental group using BumptUp mobile exercise app
- Control group (No Intervention): This group will have no access to "BumptUp" mobile exercise app and will only be provided with an educational brochure (Exercise during pregnancy)

INTERVENTIONS:
Behavioral: Experimental group using BumptUp mobile exercise app — This BumptUp app has been developed specifically for pregnancy with safety and screening feature. This intervention will be unique since the researchers will evaluate the cardiovascular health outcomes following the 8 weeks of intervention.
  Other Names: BumptUp app
  Arms: Experimental arm who will use the BumptUp mobile exercise app

SUMMARY:
The goal of this study is to determine the effectiveness of a mobile exercise app in improving cardiovascular health and motivation to exercise in pregnant women who are healthy, in their 2nd trimester, between 18-45 years age, and do not do exercise currently. The aims of this study are determine i) the effect of a mobile app (BumptUp) to increase motivation to exercise as assessed by questionnaire, and ii) the changes may occur in cardiovascular health outcomes such as increased percent Flow-Mediated Dilation (FMD), Heart Rate Variability (HRV), and decreased Pulse Wave Velocity (PWV) over an 8-week period of intervention. Researchers will compare this to pregnant women who are healthy, in their 2nd trimester, between 18-45 years age, and who will not be using the mobile app (BumptUp) for exercise. Participants who are in the experimental group will be given access to the mobile app (BumptUp) for 8 weeks. Both the control and experimental group will visit the lab for their baseline measurements (study visit 1), followed by two visits at 4 weeks (study visit 2) and 8 weeks (study visit 3) to have their heart rate variability, arterial stiffness (PWV), and vascular function (FMD) assessed. At each study visit, blood pressure, heart rate, height, and weight will also be measured. Additionally, at all three study visits, participants will fill out a questionnaire to determine motivation to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years.
* Pregnant women who are 20-24 weeks pregnant at enrollment
* Sedentary, as defined by completing less than 90 minutes of exercise each week.
* Generally healthy, uncomplicated pregnancies.
* Free of physical limitations that may interfere with alterations in daily physical activity levels.
* Single gestation.
* Have a smartphone
* Under the routine medical care of an obstetrician or certified nurse midwife during their current pregnancy.
* Women speaking English.

Exclusion Criteria:

* Physician diagnosed cardiovascular/ vascular complications (heart disease, high blood pressure, Raynaud's phenomenon etc.)
* Physician diagnosed metabolic diseases (diabetes, hypothyroidism)
* Musculoskeletal injuries (broken bones, back pain, ankle sprain, muscle pull, etc.)
* Medications that may impact blood vessel function such as hypertension medication (Angiotensin converting enzyme inhibitor, Angiotensin receptor blocker, Calcium channel blocker, beta blocker), lipid lowering agents (statins), Nitrates, steroids, etc.
* Complications associated with pregnancy that would be exacerbated by exercise such as lung disease, persistent spotting/bleeding or Placental Previa, premature labor, ruptured membranes, evidence of intrauterine growth restriction, pregnancy induced hypertension or pre-eclampsia, uncontrolled epileptic fits/seizures.
* Smoking within the previous 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women will be recruited
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Flow mediated dilation | 8 weeks of intervention period
  The cardiovascular health via flow mediated dilation (% change from baseline) will be assessed

SECONDARY OUTCOMES:
Arterial stiffness | 8 weeks
  Cardiovascular health will be measured via arterial stiffness determining pulse wave velocity (m/sec)

OTHER OUTCOMES:
Heart rate variability | 8 weeks
  Cardiovascular health will be measured via heart rate variability (msec).
motivation to exercise | 8 weeks
  Motivation to exercise will be measured via questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No